CLINICAL TRIAL: NCT07319494
Title: Comparison of Advanced Platelet Rich Fibrin Versus Platelet Rich Fibrin as a Gap Filling Material in Immediate Implant Placement
Brief Title: Advanced PRF vs PRF for Gap Filling in Immediate Implants
Acronym: A-PRF vs PRF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Eman Magdy Ahmed, Associate Professor, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DU:024111959
Record Dates: First submitted 2025-11-30; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Comparison of Advanced Platelet-Rich Fibrin Versus Platelet-Rich Fibrin as a Gap-filling Material
Keywords: Immediate dental implant placement and socket healing
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF Group (Experimental): Participants in this arm will undergo tooth extraction followed by immediate implant placement. The extraction socket will be filled with traditional Platelet-Rich Fibrin (PRF) as the gap-filling material.
  Interventions: Procedure: Immediate dental implant and PRF
- A-PRF Group (Experimental): Participants in this arm will undergo tooth extraction followed by immediate implant placement. The extraction socket will be filled with Advanced Platelet-Rich Fibrin (A-PRF) as the gap-filling material.
  Interventions: Procedure: Immediate Dental Implant and A-PRF

INTERVENTIONS:
Procedure: Immediate Dental Implant and A-PRF — Arm 1: Advanced Platelet-Rich Fibrin (A-PRF) Participants will have a tooth extracted, the socket cleaned, and A-PRF prepared from their blood placed in the socket as a gap-filling material before immediate implant placement. Follow-up visits will assess bone and soft tissue healing and implant stability.
  Arms: A-PRF Group
Procedure: Immediate dental implant and PRF — Arm 2: Platelet-Rich Fibrin (PRF) Participants will have a tooth extracted, the socket cleaned, and traditional PRF prepared from their blood placed in the socket as a gap-filling material before immediate implant placement. Follow-up visits will assess bone and soft tissue healing and implant stability.
  Arms: PRF Group

SUMMARY:
Study type: Clinical Trial

Goal:

The goal of this clinical trial is to learn if Advanced Platelet-Rich Fibrin (A-PRF) versus traditional Platelet-Rich Fibrin (PRF) can improve bone healing and soft tissue outcomes in patients undergoing immediate dental implant placement.

Main questions it aims to answer:

Does A-PRF provide greater buccal bone preservation compared to PRF after immediate implant placement?

Does A-PRF improve soft tissue healing and reduce postoperative complications compared to PRF?

Comparison group:

Researchers will compare A-PRF to PRF as a gap-filling material in immediate implants to see if A-PRF results in better bone and soft tissue outcomes.

Participants will:

Undergo tooth extraction followed by immediate implant placement

Receive either A-PRF or PRF as the gap-filling material in the implant site

Have CBCT scans at baseline and 6 months to measure bone thickness

Have clinical assessments of soft tissue healing and implant stability

Attend follow-up visits at 1 week, 1 month, 3 months, and 6 months post-surgery

ELIGIBILITY:
Inclusion Criteria:

* The selected patients has a badly decayed mandibular posterior teeth which are indicated for extraction due to dental causes (periapical abscess, trauma or caries) not periodontal as diagnosed by periapical x-ray.
* Healthy patients who are classified according to the American Society of Anesthesiologists (ASA)(2022) physical status classification as class I.
* Patient age ≥ 20 years old.
* Surgical site with sufficient for implant placement.
* Sufficient interocclusal space for prosthesis.
* Good oral hygiene.
* Patients have thick biotype.
* Patients have socket class I.

Exclusion Criteria:

* Active periodontal diseases and periapical lesions not chronic infections.
* Patients have parafunctional
* History of alcohol or drug dependency, psychological factor that might affect the surgical or prosthodontic treatment.
* Smoking.
* Pregnant patients.
* Patients who are not willing to complete the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation | 6 month
  Implant stability will be measured by resonance frequency analysis (RFA) values expressed as implant stability quotient (ISQ) unit at 6 months post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- Delta University For Science And Technology, Al Mansurah, Egypt

DOCUMENTS (1):
  • Study Protocol (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT07319494/Prot_000.pdf